CLINICAL TRIAL: NCT03661632
Title: Phase 1/2 Study of BMS-986310 Administered Alone and in Combination With Nivolumab in Participants With Advanced Solid Tumors
Brief Title: An Investigational Immunotherapy Study of BMS-986310 Administered Alone and in Combination With Nivolumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA044-001; 2018-002108-15 (EudraCT Number)
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Part 1: BMS-986310 + Nivolumab Combination Dose Escalation
  Sub-Study A: A cohort of Cisplatin Ineligible Muscle Invasive Bladder Cancer patients will receive either monotherapy BMS-986310, or BMS-986310 + Nivolumab, or Nivolumab monotherapy.
  Sub-Study B: A cohort of PD[L]1 relapsed / refractory tumor cancer patients will be treated with monotherapy BMS-986310 followed by BMS-986310 + nivolumab
  Interventions: Drug: BMS-986310; Biological: Nivolumab
- Cohort Expansion (Experimental): Part 2: Cohort Expansion will initiate upon consideration of the totality of data from Part 1.
  BMS-986310 + Nivolumab combination will be administered in specific patient populations.
  Interventions: Drug: BMS-986310; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986310 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558

SUMMARY:
The purpose of this study is to determine if BMS-986310 administered in combination with nivolumab, will demonstrate adequate safety and tolerability, as well as a favorable risk/benefit profile, to support further clinical testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable disease per RECIST v1.1 and have at least one lesion accessible for biopsy.
* ECOG performance status less than or equal to 1

Part 1 and Sub-study B:

i) Part 1 participants must have advanced or metastatic disease where no other standard of care treatment option is possible.

ii) Sub-study B participants must have advanced or metastatic disease where no other standard of care treatment is possible, in one of the following tumor types: Renal cell carcinoma, Melanoma, colorectal cancer (CRC) microsatellite instability (MSI)-High (determined by Clinical Laboratory Improvement Amendments (CLIA) validated assay, testing methodology must be provided), Bladder cancer, Squamous Cell Carcinoma of the Head and Neck (SCCHN), and they must have had disease progression on an anti-PD-(L)1 based regimen as their most recent prior therapy

Sub-study A:

i) Participants must be newly diagnosed, no prior history of treatment for bladder cancer ii) Participants must not meet criteria for standard of care neoadjuvant therapy and must be candidates for SOC surgical resection of primary tumor.

iii) Histologically confirmed muscle-Invasive bladder cancer (MIBC) pure or mixed histology urothelial carcinoma Part 2 - Patients with relapsed / refractory solid tumors where no other standard of care treatment option is available.

Exclusion Criteria:

* History of severe adverse drug reactions to nonsteroidal anti-inflammatory drugs (NSAIDs) or Cyclooxygenase-2 (COX-2) inhibitors.
* Participants with an active, known or suspected autoimmune disease.
* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | up to 3 years
Incidence of Serious Adverse Events (SAE) | up to 3 years
Incidence of AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria | up to 3 years
Incidence of AEs leading to dose delays and discontinuation or delay in radical cystectomy (RC) | up to 3 years
Incidence of Laboratory abnormalities | up to 3 years
Incidence of death | up to 3 years

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 3 years
Median duration of response (mDOR) | up to 3 years
Progression free survival rate (PFSR) | up to 24 months
Maximum observed serum concentration (Cmax) | up to 3 years
Observed serum concentration at the end of a dosing interval (Ctau) | up to 3 years
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | up to 3 years
Apparent total body clearance (CLT/F) | up to 3 years
Area under the serum concentration-time curve in 1 dosing interval [AUC(TAU)] | up to 3 years
AUC accumulation index (AI_AUC) | up to 3 years
Cmax accumulation index (AI_Cmax) | up to 3 years
Summary changes of prostaglandin E metabolite (PGEM) in urine | up to 3 years
Summary changes of tumor necrosis factor (TNFa) in blood | up to 3 years
Summary of PK parameters at T-HALF | up to 3 years
Summary of PK parameter AUC(INF) after single dose | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (4):
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Ghent
- Local Institution, Toronto, Ontario, Canada

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm